CLINICAL TRIAL: NCT00001849
Title: New Imaging Modalities in the Evaluation of Patients With Ectopic Cushing's Syndrome
Brief Title: New Imaging Techniques in the Evaluation of Patients With Ectopic Cushing Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 990055; 99-CH-0055 (Other: National Institutes of Health (NIH) Clinical Center)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-01

CONDITIONS: Cushing Syndrome; Endocrine Disease
Keywords: PET; fluorine -18(18F)-DOPA; Pentetreotide; ACTH; Octreotide; Cushing's Syndrome; Ectopic Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome; Endocrine System Diseases | interventions — pentetreotide; fluorodopa F 18; Tomography, X-Ray Computed; Magnetic Resonance Imaging; Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Comparison of results in patients receiving similar imaging scans
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Cushing Syndrome (Experimental): Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Interventions: Drug: Pentetreotide; Drug: 18F-DOPA; Device: CT scan; Device: MRI; Drug: 18-FDG

INTERVENTIONS:
Drug: Pentetreotide — Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the conventional dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
  Other Names: [111In-diethylenetriaminepentaacetic acid-D-Phe]-pentetreotide
Drug: 18F-DOPA — 18F-DOPA is a radiolabeled amino acid used as a radiotracer in positron emission tomography (PET). Limited to 3 doses over the course of the study.
  Other Names: 6-fluoro-L-DOPA; 56494
Device: CT scan — CT scan of chest, abdomen, neck and /or pelvis
  Other Names: computed tomography scan
Device: MRI — MRI scan of head/pituitary, chest, abdomen, neck and /or pelvis
  Other Names: magnetic resonance imaging scan
Drug: 18-FDG — FDG PET scan of body
  Other Names: 18-fluorine fluorodeoxyglucose PET scan

SUMMARY:
Cushing Syndrome is an endocrine disorder causing an over production of the hormone cortisol. Cortisol is produced in the adrenal gland as a response to the production of corticotropin (ACTH) in the pituitary gland.

Between 10% and 20% of patients with hypercortisolism (Cushing Syndrome) have ectopic production of the hormone ACTH. Meaning, the hormone is not being released from the normal site, the pituitary gland. In many cases the ectopic ACTH is being produced by a tumor of the lung, thymus, or pancreas. However, in approximately 50% of these patients the source of the ACTH cannot be found even with the use of extensive imaging studies such as computed tomography (CT) scans, magnetic resonance imaging (MRI), and nuclear scans (111-indium pentetreotide). The ability of these tests to locate the source of the hormone production is dependent on the changes of anatomy and / or the dose and adequate uptake of the radioactive agent. The inability to detect the source of ectopic ACTH production often results in unnecessary pituitary surgery or irradiation.

Unlike the previously described tests, positron emission tomography (PET scan) has the ability to detect pathologic tissue based on physiologic and biochemical processes within the abnormal tissue.

This study will test whether fluorine-18-fluorodeoxyglucose (FDG), fluorine-18-dihydroxyphenylalanine (F-DOPA) or use of a higher dose of 111-indium pentetreotide can be used to successfully localize the source of ectopic ACTH production.

DETAILED DESCRIPTION:
Between 10 percent and 20 percent of patients with hypercortisolism (Cushing syndrome) have ectopic production of adrenocorticotropin hormone (ACTH) that causes cortisol excess. In approximately 50 percent of these patients, the source of ACTH cannot be found despite very detailed and extensive examination including imaging studies such as computed tomography scanning, magnetic resonance imaging, and octreotide scan (octreoscan) using the conventional low dose of indium-111 pentetreotide. The sensitivity and specificity of these imaging studies depends on anatomic alterations and/or the dose and adequate uptake of radiopharmaceutical. In contrast, positron emission tomography (PET) has the ability to detect pathologic tissue based on physiologic and biochemical processes within the abnormal tissue. This protocol tests whether fluorine-18 dihydroxyphenylalanine (F-DOPA) or use of a higher dose of indium-111 pentetreotide (Octreoscan) can be used to localize successfully the source of ectopic ACTH production. In addition the study examines whether administration of the glucocorticoid antagonist mifepristone can improved the sensitivity of the standard dose Octreoscan. Eligible patients participating in this arm of the study will have a second standard dose scan. Others will receive a higher dose octreoscan instead.

ELIGIBILITY:
* INCLUSION CRITERIA:

All eligible patients are invited to participate in this protocol. Patients are adults with possible ectopic Cushing syndrome. Since both men and women are affected with ectopic Cushing syndrome, both sexes are studied. All ethnic and racial groups are at risk and will be included. Patients must be willing to return to the National Institutes of Health (NIH) Clinical Center for follow-up studies.

EXCLUSION CRITERIA:

Pregnant or lactating women. A pregnancy test is performed in women of childbearing potential (up to age 55) unless they have a history of hysterectomy.

Children (age less than18) are excluded. Because ectopic ACTH secretion is rare in this age group, the likelihood of benefit is less and does not balance the risk of radiation.

Patients taking medications that alter CYP3A4 activity will not be eligible for the mifepristone study, since this P450 system metabolizes mifepristone. Such participants would receive a clinical high dose (18 mCi) octreoscan (H-OCT) instead, if the standard 6 mCi octreoscan (L-OCT) was negative. Patients with hypokalemia (K < 3.5 milliequivalent (mEq)/L) despite medical therapy with replacement or mineralocorticoid antagonists will also be excluded from the mifepristone studies.

The presence of:

* severe active infection.
* clinically significantly impaired cardiovascular (e.g., history of abnormally low ejection fraction, the presence of moderate pulmonary fluid overload or leg edema, and blood pressure over 190/100), abnormal coagulation (partial thromboplastin time or prothrombin time elevated by 30 percent above the normal values), hematopoietic (hematocrit less than 30 percent, hemoglobin below 10 g/dl, white count below 3000 K/microliter (UL), and platelets below 100,000 K/mm(3)), hepatic (liver enzymes elevated by 3-fold above normal values) or renal function (plasma creatinine level over 2.0).
* impaired mental capacity or markedly abnormal psychiatric evaluation that precludes informed consent.
* body weight over 136 kg, which is the limit for the tables used in the scanning areas.
* combined blood withdrawal, during the six weeks preceding the study, of greater than 450 ml.
* known allergy to 111-indium pentetreotide or other somatostatin analogues.
* strong evidence for Cushing disease. This includes those with positive inferior petrosal sinus sampling or a lesion on pituitary MRI.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 1999-05-20 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Findling JW, Tyrrell JB. Occult ectopic secretion of corticotropin. Arch Intern Med. 1986 May;146(5):929-33. PMID 3963984
- [Background] Jex RK, van Heerden JA, Carpenter PC, Grant CS. Ectopic ACTH syndrome. Diagnostic and therapeutic aspects. Am J Surg. 1985 Feb;149(2):276-82. doi: 10.1016/s0002-9610(85)80085-4. PMID 2982290
- [Background] Trainer PJ, Grossman A. The diagnosis and differential diagnosis of Cushing's syndrome. Clin Endocrinol (Oxf). 1991 Apr;34(4):317-30. doi: 10.1111/j.1365-2265.1991.tb03773.x. No abstract available. PMID 1879062
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-CH-0055.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on physician referral to the NIH Clinical Center from 4/1999 to 12/2015. The first participant enrolled on 5/20/99 and the last participant enrolled on 11/19/15. Of 95 enrolled participants, 68 met inclusion criteria and underwent imaging studies.
Pre-assignment Details: 27 patients had biochemical testing consistent with Cushing's disease and were excluded from additional participation.
Units Other Than Participants: lesions, total body
Groups:
- Patients With Presumed Ectopic ACTH Secretion: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Pentetreotide: Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the conventional dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
  FDG-PET: Fluorodeoxyglucose (FDG) is a radiolabeled glucose used as a radiotracer in positron emission tomography (PET); FDG-PET was deleted as a required research study in 2004; thereafter used as clinically indicated.
  Fluorine-18 dihydroxyphenylalanine (F-DOPA) is a radiolabeled amino acid used as a radiotracer in positron emission tomography. F-DOPA scans are limited to 3 over the course of the study.
  CT Scans, MRI scans
Period: Overall Study
Arm/Group | Patients With Presumed Ectopic ACTH Secretion
Started | 68; 68 lesions, total body
Completed | 54; 54 lesions, total body (Patients completed when an ectopic ACTH-secreting tumor was identified)
Not Completed | 14; 14 lesions, total body
Not completed — Death | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — tumor remained occult | 6

BASELINE CHARACTERISTICS:
Groups:
- Patients With Presumed Ectopic ACTH Secretion: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Pentetreotide: Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the conventional dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
  FDG-PET: FDG is a radiolabeled glucose used as a radiotracer in positron emission tomography; FDG-PET deleted as required research study in 2004; thereafter used as clinically indicated.
  Fluorine-18 (18F)-DOPA: 18F-DOPA is a radiolabeled amino acid used as a radiotracer in positron emission tomography. F-DOPA scans are limited to 3 over the course of the study.
  CT Scans, MRI scans
Arm/Group | Patients With Presumed Ectopic ACTH Secretion
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 53
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 68
Participants with presumed ectopic corticotropin (ACTH) syndrome [Count of Participants; unit: Participants] | 68

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Imaging Modalities for the Detection of ACTH-secreting Non-pituitary Tumor in Patients
Description: The percentage of patients in whom imaging correctly identified an ACTH-secreting non-pituitary tumor within six months of resection or in which imaging identified a recurrence at a site of previous resection.
Time Frame: six months or less
Population: Tumors identified by specific imaging modality in each patient
Measure: Number (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: lesions on imaging
Groups:
- CT Scan Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  CT Scans of chest, abdomen, neck and/or pelvis are used.
- Magnetic Resonance Imaging (MRI) Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  MRI scans of chest, abdomen, neck, head, and/or pelvis obtained at 1.5 Tesla are shown.
- Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  FDG-PET: FDG is a radiolabeled glucose used as a radiotracer in; FDG-PET deleted as required research study in 2004; thereafter used as clinically indicated.
- [18F]-L-3,4-dihydroxyphenylalanine (18F-DOPA) PET Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  18F-DOPA: F-DOPA is a radiolabeled amino acid used as a radiotracer in positron emission tomography. F-DOPA scans are limited to 3 over the course of the study.
- Standard Dose Pentetreotide Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Pentetreotide: Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the standard dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
- High Dose (18 mCi) Pentetreotide Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Pentetreotide: Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the conventional dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
Arm/Group | CT Scan Results | Magnetic Resonance Imaging (MRI) Results | Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Results | [18F]-L-3,4-dihydroxyphenylalanine (18F-DOPA) PET Results | Standard Dose Pentetreotide Results | High Dose (18 mCi) Pentetreotide Results
Number analyzed (Participants) | 54 | 48 | 9 | 23 | 51 | 21
Number analyzed (lesions on imaging) | 69 | 55 | 13 | 24 | 57 | 22
percentage of patients | 96.3 [87.7 to 99.0] | 77.1 [61.2 to 85.1] | 66.7 [35.4 to 87.9] | 100 [85.7 to 100] | 45.1 [32.3 to 58.6] | 42.9 [24.5 to 63.5]

2. Primary Outcome: Sensitivity of Imaging Modalities for the Detection of ACTH-secreting Non-pituitary Tumor in Specific Lesions
Description: The percentage of lesions for which imaging correctly identified an ACTH-secreting non-pituitary tumor within six months of resection or for which imaging identified a recurrence at a site of previous resection.
Time Frame: six months or less
Population: Tumors identified by specific imaging modality by lesions
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions on imaging
Groups:
- MRI Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  MRI scans of chest, abdomen, neck, head, and/or pelvis obtained at 1.5 Tesla are shown.
- FDG-PET Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  FDG-PET: FDG is a radiolabeled glucose used as a radiotracer in positron emission tomography; FDG-PET deleted as required research study in 2004; thereafter used as clinically indicated.
- F-DOPA PET Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  18F-DOPA: F-DOPA is a radiolabeled amino acid used as a radiotracer in positron emission tomography. F-DOPA scans are limited to 3 over the course of the study.
- High Dose (18 mCi) Octreotide Results: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Pentetreotide: Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the conventional dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
Arm/Group | CT Scan Results | MRI Results | FDG-PET Results | F-DOPA PET Results | Standard Dose Pentetreotide Results | High Dose (18 mCi) Octreotide Results
Number analyzed (Participants) | 54 | 48 | 9 | 23 | 51 | 21
Number analyzed (lesions on imaging) | 69 | 55 | 13 | 24 | 57 | 22
percentage of lesions | 75.4 [64 to 84] | 67.3 [53.4 to 77.8] | 46.2 [23.2 to 71] | 95.8 [79.8 to 99.3] | 40.4 [28.6 to 53.3] | 40.9 [23.3 to 61.3]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored during each inpatient admission, generally 7 - 14 days.
Description: AEs within 24 hrs of F-DOPA (ten half-lives rounded up), would be reported to the sponsor. Minor deviations in standard care, such as decisions not to schedule all possible imaging (eg deleting pelvic scans in a patient with a lung mass) will not be reported. Expected AEs (those in the protocol/F-DOPA investigator's brochure, and thromboembolism, hypertension, infection, metabolic derangements, which are common in Cushing's syndrome) would be reported only if they become unanticipated problems.
Groups:
- Patients With Cushing Syndrome: Patients receive various types of radiologic or nuclear medicine scans to identify tumor
  Pentetreotide: Binds primarily to the somatostatin receptors subtypes (sst) 2 and 5. A high dose (18mCi) was used if the conventional dose (6mCi) was negative and scheduling was available. High doses limited to 3 over the course of the study.
  18F-DOPA: F-DOPA is a radiolabeled amino acid used as a radiotracer in positron emission tomography. Limited to 3 doses over the course of the study.
  CT scan: CT scan of chest, abdomen, neck and /or pelvis
  MRI: MRI scan of head/pituitary, chest, abdomen, neck and /or pelvis
  18-FDG: FDG PET scan of body
Arm/Group | Patients With Cushing Syndrome
All-Cause Mortality (participants affected / at risk) | 4/68
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

LIMITATIONS AND CAVEATS:
Small number of subjects with this rare disorder; radiation safety risk limited number of some scans; difficulty in scheduling all scans due to lack of availability of slots or radionuclide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT00001849/Prot_SAP_000.pdf